CLINICAL TRIAL: NCT01816893
Title: Hypoglycemia and Autonomic Nervous System Function
Acronym: HypoANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Gail Adler, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2004P001233; R01DK063296 (NIH); M01RR002635 (NIH)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Results first posted 2018-03-06 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Autonomic Nervous System; baroreflex sensitivity; muscle sympathetic nerve activity; lower body negative pressure
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euglycemic hyperinsulinemic clamp (Sham Comparator): participant undergoes a euglycemic hyperinsulinemic clamp
  Interventions: Other: Euglycemic hyperinsulinemic clamp
- Hypoglycemic hyperinsulinemic clamp (Active Comparator): participant undergoes a hypoglycemic hyperinsulinemic clamp
  Interventions: Other: Hypoglycemic hyperinsulinemic clamp

INTERVENTIONS:
Other: Hypoglycemic hyperinsulinemic clamp
  Arms: Hypoglycemic hyperinsulinemic clamp
Other: Euglycemic hyperinsulinemic clamp
  Arms: Euglycemic hyperinsulinemic clamp

SUMMARY:
The goals of this proposal are to determine the effects of hypoglycemia on the autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria

* Healthy volunteers
* Males and females age 18 to 50 years

Exclusion Criteria

* Pregnancy
* Lactation
* Subjects who smoke or are on other forms of nicotine will be excluded
* Clinically evident coronary artery, cerebrovascular, or peripheral vascular disease, or presence of systemic illness that might affect autonomic function. Such illnesses include diabetes mellitus, congestive heart failure, hypertension, renal, pulmonary, hepatic disease, anemia, malignancies, untreated thyroid disease, and alcoholism.
* Current major depressive illness
* Any individuals on oral, injected, inhaled or topical corticosteroids within the last year or oral contraceptives within the past 3 months will be excluded.
* Use of medications other than thyroxine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2004-06-08 (Actual); Primary Completion 2007-11-06 (Actual); Study Completion 2007-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital; Roy L Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
The data collected will comply with the NIH requirements for timely release and data sharing. Data will be shared in the form of publications and presentations in scientific forums. As the NIH has noted, the investigators reserve the right to keep the data restricted in order to perform the initial analyses for this grant proposal and will continue to use the data for further, but not prolonged, exclusive use. Of note, the sharing of this data will be limited by at least the following issues, some unique to this proposal and some not unique. Some of the data obtained in this study is defined to be sensitive in nature, which may restrict its ability to be shared. Data may only be shared with the approval of our IRB and is limited by HIPPA and any other regulations that may be promulgated during the course of this proposal.

REFERENCES:
- [Result] Dotson S, Freeman R, Failing HJ, Adler GK. Hypoglycemia increases serum interleukin-6 levels in healthy men and women. Diabetes Care. 2008 Jun;31(6):1222-3. doi: 10.2337/dc07-2243. Epub 2008 Mar 10. PMID 18332163
- [Result] Adler GK, Bonyhay I, Failing H, Waring E, Dotson S, Freeman R. Antecedent hypoglycemia impairs autonomic cardiovascular function: implications for rigorous glycemic control. Diabetes. 2009 Feb;58(2):360-6. doi: 10.2337/db08-1153. Epub 2008 Dec 3. PMID 19056608
- [Result] Gibbons CH, Adler GK, Bonyhay I, Freeman R. Experimental hypoglycemia is a human model of stress-induced hyperalgesia. Pain. 2012 Nov;153(11):2204-2209. doi: 10.1016/j.pain.2012.06.030. Epub 2012 Aug 23. PMID 22921261
- [Result] Adler GK, Bonyhay I, Curren V, Waring E, Freeman R. Hypoglycaemia increases aldosterone in a dose-dependent fashion. Diabet Med. 2010 Nov;27(11):1250-5. doi: 10.1111/j.1464-5491.2010.03087.x. PMID 20950382

RESULTS

PARTICIPANT FLOW:
Groups:
- Euglycemic Clamp/ Washout Period/ Hypoglycemic Clamp: 1. Participant undergoes a euglycemic hyperinsulinemic clamp
  2. Participant undergoes a 1-3 month washout period
  3. Participant undergoes a hypoglycemic hyperinsulinemic clamp
- Hypoglycemic Clamp/ Washout Period/ Euglycemic Clamp: 1. Participant undergoes a hypoglycemic hyperinsulinemic clamp
  2. Participant undergoes a 1-3 month washout period
  3. Participant undergoes a euglycemic hyperinsulinemic clamp
Period: Euglycemic Clamp/ Hypoglycemic Clamp
Arm/Group | Euglycemic Clamp/ Washout Period/ Hypoglycemic Clamp | Hypoglycemic Clamp/ Washout Period/ Euglycemic Clamp
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Euglycemic Clamp/ Washout Period/ Hypoglycemic Clamp | Hypoglycemic Clamp/ Washout Period/ Euglycemic Clamp
Started | 11 | 11
Completed | 9 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Hypoglycemic Clamp/ Euglycemic Clamp
Arm/Group | Euglycemic Clamp/ Washout Period/ Hypoglycemic Clamp | Hypoglycemic Clamp/ Washout Period/ Euglycemic Clamp
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Euglycemic Clamp/ Washout Period/ Hypoglycemic Clamp | Hypoglycemic Clamp/ Washout Period/ Euglycemic Clamp | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 29 (8) | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 6 | 9 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Baroreflex Sensitivity
Description: The change in baroreflex sensitivity (milliseconds/mm Hg) is calculated as baroreflex sensitivity (milliseconds/mm Hg) on day 3 [assessed 16 hours after the clamp] minus baroreflex sensitivity (milliseconds/mm Hg) on day 1 [baseline assessment on the day prior to the clamp]). Change in baroreflex sensitivity in euglycemic clamp arm is compared to change in baroreflex sensitivity in hypoglycemic arm.
Time Frame: 16 hours after euglycemic and hypoglycemic clamps as compared to baseline
Population: 20 subjects completed both arms, but only 18 had the change in BRS outcome for both arms.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Groups:
- Euglycemic Clamp: participant undergoes a euglycemic hyperinsulinemic clamp
  Euglycemia
- Hypoglycemic Clamp: participant undergoes a hypoglycemic hyperinsulinemic clamp
  Hypoglycemia
Arm/Group | Euglycemic Clamp | Hypoglycemic Clamp
Number analyzed (Participants) | 18 | 18
ms/mmHg | 2.3 (6.3) | -1.6 (4.3)

2. Secondary Outcome: Muscle Sympathetic Nerve Activity
Description: Muscle sympathetic nerve activity (MSNA), at rest and immediately after nitroprusside, was measured on Day 3 about 16 hours after the euglycemic and hypoglycemic clamps.
Time Frame: 16 hours after euglycemic and hypoglycemic clamps
Population: 20 subjects completed both arms, but only 5 had the muscle sympathetic nerve activity outcome for both arms.
Measure: Mean (Standard Deviation); unit: bursts/ minute
Arm/Group | Euglycemic Clamp | Hypoglycemic Clamp
Number analyzed (Participants) | 5 | 5
bursts/ minute
  At rest | 33.64 (3.3) | 26.4 (4.8)
  With Nitroprusside | 53.4 (3.7) | 40.1 (2.7)

3. Secondary Outcome: Catecholamine Response to Lower-body Negative Pressure
Description: Plasma norepinephrine response to lower body negative pressure (at the minus 40 mm Hg data point) on Day 3 about 16 to 20 hours after completion of the euglycemic or hypoglycemic clamp.
Time Frame: 16 hours after euglycemic and hypoglycemic clamps
Population: Of the 22 subjects who started the protocol, 20 completed both arms.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Euglycemic Clamp | Hypoglycemic Clamp
Number analyzed (Participants) | 20 | 20
nmol/L | 3.0 (0.3) | 2.0 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for about a week (during each 3-day assessment and for a few days afterwards).
Groups:
- Euglycemic Clamp: Participant undergoes a euglycemic hyperinsulinemic clamp
- Hypoglycemic Clamp: Participant undergoes a hypoglycemic hyperinsulinemic clamp
Arm/Group | Euglycemic Clamp | Hypoglycemic Clamp
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No